CLINICAL TRIAL: NCT01763541
Title: Gonadal Steroid Regulation of the Natriuretic Peptide System
Brief Title: Study of the Effect of Testosterone and Estradiol on NP Responses to Acute and Chronic Salt Loading
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Director, Neuroendocrine Research Program in Women's Health, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012P002337
Record Dates: First submitted 2012-11-13; First posted 2013-01-09 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
Keywords: Natriuretic Peptides
MeSH Terms: conditions — Hypertension | interventions — Leuprolide; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone (Other): To determine the effect of testosterone on the NP responses to acute and chronic salt loading.
  One testosterone patch (Androderm 5 mg) applied to each male subject each day for 14 days.
  Intervention: Leuprolide acetate and anastrozole
  Interventions: Drug: leuprolide acetate; Drug: Anastrozole
- Estradiol (Other): To determine the effect of estradiol on the NP responses to acute and chronic salt loading.
  Two estradiol patches (Vivelle Dot 0.1mg) will be applied to each female subject twice-a-week for 2 weeks.
  Intervention: leuprolide acetate
  Interventions: Drug: leuprolide acetate

INTERVENTIONS:
Drug: leuprolide acetate — Given to both arms to induce hypogonadism
  Other Names: Lupron Depot 3.75 mg and 7.5 mg
Drug: Anastrozole — Given to men to prevent conversion of administered testosterone to estradiol.
  Other Names: Arimidex
  Arms: Testosterone

SUMMARY:
There is gender dimorphism in cardiovascular risk, with men at higher risk than women. However, the fundamental basis for the protective effect of female sex remains unclear. Recent data implicate the natriuretic peptide (NP) system as an important determinant of blood pressure. Also, NP levels are twice as high in women of reproductive age than in men, and gonadal steroids are important determinants of circulating NPs. These are the marked, but poorly understood differences in the NP status between men and women. The investigators hypothesize that gonadal steroids regulate NP release, specifically that testosterone inhibits and estrogen activates the NP axis, leading to differences in both resting NP levels and dynamic responses of the NP, RAAS, and kidneys to acute and chronic salt loading. Understanding the basis for gender differences in NP function should provide important insights regarding mechanisms underlying hypertension in men versus women.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* no history of hypertension
* normal BMI
* Male: normal testosterone and free testosterone levels
* Female: regular menses, negative pregnancy test, no sex steroid therapy >/=3 mos

Exclusion Criteria:

* on hypertensives, diuretics, or insulin
* with diabetes mellitus
* estimated creatinine clearance <60 ml/min
* prior cardiovascular, liver or renal disease
* history of hormonally-responsive cancer
* elevated liver function test (LFTs)
* atrial fibrillation
* abnormal sodium or potassium levels
* taking medications that directly impact the endocrine system (exogenous hormones, steroids, etc.)
* taking medications that indirectly impact the endocrine system (SSRIs, opioids, finasteride, etc.)
* with untreated hyper- or hypothyroidism
* smoker
* psychiatric history
* Women: not willing to abstain from getting pregnant during the course of the study, with abnormal menstrual cycle, or who have osteoporosis
* Men: with polycythemia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
NP levels in men with testosterone patch and low-salt diet | At day 7 of week of testosterone administration with low-salt diet
  B-type natriuretic peptide (BNP), Atrial natriuretic peptide (ANP), amino-terminal brain natiuretic peptide (N-BNP), amino-terminal atrial natiuretic peptide (N-ANP), cyclic guanosine monophosphate (cGMP)
NP levels in men with testosterone patch and high-salt diet | At day 7 of week of testosterone administration with high-salt diet
  B-type natriuretic peptide (BNP), Atrial natriuretic peptide (ANP), amino-terminal brain natiuretic peptide (N-BNP), amino-terminal atrial natiuretic peptide (N-ANP), cyclic guanosine monophosphate (cGMP)
NP levels in women with estradiol patch and low-salt diet | At day 7 of week of estradiol administration with low-salt diet
  B-type natriuretic peptide (BNP), Atrial natriuretic peptide (ANP), amino-terminal brain natiuretic peptide (N-BNP), amino-terminal atrial natiuretic peptide (N-ANP), cyclic guanosine monophosphate (cGMP)
NP levels in women with estradiol patch and high-salt diet | At day 7 of week of estradiol administration with high-salt diet
  B-type natriuretic peptide (BNP), Atrial natriuretic peptide (ANP), amino-terminal brain natiuretic peptide (N-BNP), amino-terminal atrial natiuretic peptide (N-ANP), cyclic guanosine monophosphate (cGMP)
NP levels in men with placebo patch and low-salt diet | At day 7 of week of placebo administration with low-salt diet
  B-type natriuretic peptide (BNP), Atrial natriuretic peptide (ANP), amino-terminal brain natiuretic peptide (N-BNP), amino-terminal atrial natiuretic peptide (N-ANP), cyclic guanosine monophosphate (cGMP)
NP levels in men with placebo patch and high-salt diet | At day 7 of week of placebo administration with high-salt diet
  B-type natriuretic peptide (BNP), Atrial natriuretic peptide (ANP), amino-terminal brain natiuretic peptide (N-BNP), amino-terminal atrial natiuretic peptide (N-ANP), cyclic guanosine monophosphate (cGMP)
NP levels in women with placebo patch and low-salt diet | At day 7 of week of placebo administration with low-salt diet
  B-type natriuretic peptide (BNP), Atrial natriuretic peptide (ANP), amino-terminal brain natiuretic peptide (N-BNP), amino-terminal atrial natiuretic peptide (N-ANP), cyclic guanosine monophosphate (cGMP)
NP levels in women with placebo patch and high-salt diet | At day 7 of week of placebo administration with high-salt diet
  B-type natriuretic peptide (BNP), Atrial natriuretic peptide (ANP), amino-terminal brain natiuretic peptide (N-BNP), amino-terminal atrial natiuretic peptide (N-ANP), cyclic guanosine monophosphate (cGMP)

SECONDARY OUTCOMES:
Plasma Renin Activity (PRA) levels in women on estradiol on low-salt diet | At day 7 of week of estradiol administration on low-salt diet
  Plasma Renin Activity (PRA)
Aldosterone levels in men with testosterone on low-salt diet | At day 7 of week of testosterone administration on low-salt diet
  Aldosterone
Plasma Renin Activity (PRA) levels in women on estradiol on high-salt diet | At days 6 and 7 of week of estradiol administration on high-salt diet
  Plasma Renin Activity (PRA)
Plasma Renin Activity (PRA) levels in women on placebo on low-salt diet | At day 7 of week of placebo administration on low-salt diet
  Plasma Renin Activity (PRA)
Plasma Renin Activity (PRA) levels in women on placebo on high-salt diet | At days 6 and 7 of week of placebo administration on high-salt diet
  Plasma Renin Activity (PRA)
Plasma Renin Activity (PRA) levels in men on testosterone on low-salt diet | At day 7 of week of testosterone administration on low-salt diet
Plasma Renin Activity (PRA) levels in men on testosterone on high-salt diet | At days 6 and 7 of week of testosterone administration on high-salt diet
Plasma Renin Activity (PRA) levels in men on placebo on low-salt diet | At day 7 of week of placebo administration on low-salt diet
Plasma Renin Activity (PRA) levels in men on placebo on high-salt diet | At days 6 and 7 of week of placebo administration on high-salt diet
Aldosterone levels in men on testosterone on high-salt diet | At days 6 and 7 of week of testosterone administration on high-salt diet
Aldosterone levels in men on placebo on high-salt diet | At days 6 and 7 of week of placebo administration on high-salt diet
Aldosterone levels in men on placebo on low-salt diet | At day 7 of week of placebo administration on low-salt diet
Aldosterone levels in women on estradiol on high-salt diet | At days 6 and 7 of week of estradiol administration on high-salt diet
Aldosterone levels in women on estradiol on low-salt diet | At day 7 of week of estradiol administration on low-salt diet
Aldosterone levels in women on placebo on high-salt diet | At days 6 and 7 of week of placebo administration on high-salt diet
Aldosterone levels in women on placebo on low-salt diet | At day 7 of week of placebo administration on low-salt diet
Urinary sodium concentration in women on estradiol on high-salt diet | 0, 60, and 120 minute of saline infusion on morning of day 7 of estradiol administration on high-salt diet
Urinary sodium concentration in women on placebo on high-salt diet | 0, 60, and 120 minute of saline infusion on morning of day 7 of placebo administration on high-salt diet
Urinary sodium concentration in men on testosterone on high-salt diet | 0, 60, and 120 minute of saline infusion on morning of day 7 of testosterone administration on high-salt diet
Urinary sodium concentration in men on placebo on high-salt diet | 0, 60, and 120 minute of saline infusion on morning of day 7 of placebo administration on high-salt diet

CONTACTS AND LOCATIONS:
Overall Officials: Karen Miller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States